CLINICAL TRIAL: NCT05451537
Title: Correlation of Formyl Peptide Receptor 1 With Sepsis-related Encephalopathy: A Prospective Cohort Study
Brief Title: Correlation of Formyl Peptide Receptor 1 With Sepsis-related Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-2022-0139
Record Dates: First submitted 2022-06-23; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-06

CONDITIONS: Sepsis-Associated Encephalopathy
MeSH Terms: conditions — Sepsis-Associated Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis associated encephalopathy group: Patients were diagnosed with sepsis related encephalopathy
- None sepsis associated encephalopathy group: Patients were not diagnosed with sepsis related encephalopathy

SUMMARY:
The pathogenesis of sepsis-associated encephalopathy (SAE) is unclear, Formylpeptide receptor 1 (FPR1) is a cell membrane receptor that recruits leukocytes and mediates inflammatory responses after activation, but its role and mechanism in SAE are unknown. This project intends to clarify the relationship between FPR1 activation and SAE from the clinical. The investigators enrolled 100 patients with sepsis in ICU. Patients were divided into two groups according to diagnostic criteria: SAE group and none-SAE group. Whole blood was collected. The serum FPR1 protein level was measured using a commercial enzyme-linked immunosorbent assay. After whole blood RNA was extracted, the expressions of FPR1 and a reference gene were quantified by an automated one-step Taqman RT-PCR assay. Multiple logistical regression analysis was used to identify the independent factors (including FPR1 activation) for the prediction of SAE outcomes.

DETAILED DESCRIPTION:
Background The pathogenesis of sepsis-associated encephalopathy (SAE) is unclear, and there are no desired therapeutic methods. Formylpeptide receptor 1 (FPR1) is a cell membrane receptor that recruits leukocytes and mediates inflammatory responses after activation, but its role and mechanism in SAE are unknown. Our previous studies have shown that the expression of FPR1 in the hippocampus of septic mice is increased; FPR1 knockout reduces mortality and microglial activation. Based on this, it is hypothesized that during sepsis, FPR1 induces the migration and recruitment of neutrophils and monocytes to the brain, at the same time, FPR1 activation of microglia mediates brain inflammatory response and cell death, these factors induces or aggravates cognitive dysfunction. This project intends to clarify the relationship between FPR1 activation and SAE from the clinical. The study will provide some useful data for the mechanism study of SAE.

Methods Inclusion criteria for participants were patients with an age of 18-70 years and an inclusion within 24 hours after the beginning of severe sepsis or septic shock according to the criteria that were established by the international guidelines for management of severe sepsis and septic shock.

Patients were excluded from the study if they had a previous diagnosis of a neuropsychiatric disease (head trauma, cerebral stroke, epilepsy, and intracranial infection), current brain disorders (hepatic encephalopathy, pulmonary encephalopathy, and severe electrolyte imbalance), concurrent hematologic diseases, malignant tumor, postcardiac arrest, or melanoma or if they were undergoing cancer chemotherapy.

Demographic, clinical, and laboratory data were retrieved after intensive care unit (ICU) admission from the medical records made by two physicians. Age, gender, Acute Physiology and Chronic Health Evaluation II score (APACHE II score), Sequential Organ Failure Assessment (SOFA) score, GCS score, and infection sites were collected and determined during the first 24 hours of admission. basic laboratory tests, including blood lactate, B-type natriuretic peptide, and inflammatory markers of white blood cell count (WBC), procalcitonin (PCT), and C-reactive protein (CRP), were detected on admission. The GCS and mental status of the patients were evaluated twice a day, at eight o'clock in the morning and six o'clock in the afternoon, including SAE symptoms of somnolence, stupor, coma, confusion, disorientation, agitation, irritability, and decreased level of GCS. Sepsis-associated encephalopathy (SAE) was defined as cerebral dysfunction in the presence of severe sepsis as well as the presentation of two or more of the symptoms listed above after complete withdrawal of sedation.

Original cerebral dysfunction derived from hypoxic encephalopathy, severe hypoglycemia, intracranial hemorrhage, epilepsy relapse, acute ischemic stroke, and hyponatremia were excluded. Supportive treatments, such as the use of a ventilator, length of ICU stay, and 28-day mortality, were also included for assessment.

Blood samples were collected from patients on admission through venipuncture. the resultant serum samples were aliquoted and stored at -80°C until further analysis. The serum FPR1 protein level was measured using a commercial enzyme-linked immunosorbent assay.

Patients were divided into two groups according to diagnostic criteria: SAE group and none SAE group. Whole blood was collected. The serum FPR1 protein level was measured using a commercial enzyme-linked immunosorbent assay. After whole blood RNA was extracted, the expressions of FPR1 and a reference gene were quantified by an automated one-step Taqman RT-PCR assay.

Multiple logistical regression analysis was used to identify the independent factors for the prediction of SAE outcomes using the forward stepwise method with the likelihood ratio test. Correlations between variables were tested by the Pearson linear regression test. Receiver operating characteristics (ROC) analysis was used to qualify marker performance, and ROC curves were constructed to assess the sensitivity, specificity, and respective areas under the curves (AUCs) of the FPR1 protein performance with 95% CI. A value of P<0.05 was considered statistically significant.

The primary outcome is the comparison of FPR1 levels in patients with and without sepsis related encephalopathy. Secondary Outcome Measures: the comparison of laboratory data, inflammatory cytokines levels in patients with and without sepsis related encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for participants were patients with an age of 18-70 years and an inclusion within 24 hours after the beginning of severe sepsis or septic shock according to the criteria that were established by the international guidelines for management of severe sepsis and septic shock.

Exclusion Criteria:

* Patients were excluded from the study if they had a previous diagnosis of a neuropsychiatric disease (head trauma, cerebral stroke, epilepsy, and intracranial infection), current brain disorders (hepatic encephalopathy, pulmonary encephalopathy, and severe electrolyte imbalance), concurrent hematologic diseases, malignant tumor, postcardiac arrest, or melanoma or if they were undergoing cancer chemotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe sepsis and septic shock, Sepsis associated encephalopathy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
The comparison of FPR1 levels in patients with and without sepsis related encephalopathy | 3 days
  The comparison of serum FPR1 protein levels (ng/ml) in patients with and without sepsis related encephalopathy

SECONDARY OUTCOMES:
The comparison of Inflammatory cytokines levels in patients with and without sepsis related encephalopathy | 3 days
  The comparison of serum IL-1β and IL-6 concentrations (ng/ml) in patients with and without sepsis related encephalopathy
The comparison of peripheral blood leukocytes in patients with and without sepsis related encephalopathy | 3 days
  The comparison of peripheral blood leukocytes count in patients with and without sepsis related encephalopathy
The comparison of S-100β levels in patients with and without sepsis related encephalopathy | 3 days
  The comparison of peripheral blood S-100β protein concentrations (ng/ml) in patients with and without sepsis related encephalopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China